CLINICAL TRIAL: NCT00531154
Title: Evaluation of the Dental Health Condition in Obesity Patients Before and After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: heling-HMO-CTIL
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Obesity; Periodontitis; Caries; Periapical Lesion
MeSH Terms: conditions — Obesity; Periodontitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aim of this study is to investigate whether there was an association between obesity and periodontitis, tendency to caries and periapical lesions.

People who have a higher body mass index produce cytokines (hormone-like proteins), that lead to systemic/chronic inflammation (like periodontitis and periapical lesions), and obesity related dietary habits could result in an increment of dental caries because both the amount and the frequency of sucrose ingestion are important factors associated with the aetiology of the oral disease.

ELIGIBILITY:
Inclusion Criteria:

* Obese pateints who intended to go bariatric surgery.

Exclusion Criteria:

* Coronary heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Heling, Prof., Principal Investigator
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Pischon N, Heng N, Bernimoulin JP, Kleber BM, Willich SN, Pischon T. Obesity, inflammation, and periodontal disease. J Dent Res. 2007 May;86(5):400-9. doi: 10.1177/154405910708600503. PMID 17452558
- [Background] Linden G, Patterson C, Evans A, Kee F. Obesity and periodontitis in 60-70-year-old men. J Clin Periodontol. 2007 Jun;34(6):461-6. doi: 10.1111/j.1600-051X.2007.01075.x. Epub 2007 Apr 2. PMID 17403015
- [Background] Karjalainen S. Eating patterns, diet and dental caries. Dent Update. 2007 Jun;34(5):295-8, 300. doi: 10.12968/denu.2007.34.5.295. PMID 17624146
- [Result] Heling I, Sgan-Cohen HD, Itzhaki M, Beglaibter N, Avrutis O, Gimmon Z. Dental complications following gastric restrictive bariatric surgery. Obes Surg. 2006 Sep;16(9):1131-4. doi: 10.1381/096089206778392211. PMID 16989694